CLINICAL TRIAL: NCT06999278
Title: LIGHT - Levothyroxine for Isolated Gestational HypoThyroidism in Women With Recurrent Pregnancy Loss: a Multicenter Randomized, Double-blind, Placebo-controlled Trial - a Study Protocol
Brief Title: LIGHT Trial: Levothyroxine for Gestational Hypothyroidism in Recurrent Pregnancy Loss
Acronym: LIGHT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Qiong Luo, Prof., Women's Hospital School Of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-20250069-R
Record Dates: First submitted 2025-03-19; First posted 2025-05-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Abortion, Habitual
Keywords: recurrent pregnancy loss; isolated maternal hypothyroidism; levothyroxine; adverse pregnancy outcomes; live birth; neonatal complications
MeSH Terms: conditions — Abortion, Habitual | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and Investigators Both participants and investigators are blinded to the group assignments. Participants receive either levothyroxine (50 µg/day) or a placebo in identical tablets that are indistinguishable in appearance, color, shape, and weight. Investigators administering treatments and assessing outcomes remain unaware of the treatment allocation.
  Randomization and Allocation Randomization is conducted using a secure web-based system, ensuring a 1:1 allocation ratio to either the levothyroxine or placebo group. The randomization process is stratified by study centers to maintain balance across locations.
  Packaging and Labeling Study drugs, including the placebo, are packaged and labeled uniformly to prevent any visual or informational clues. Each package contains a unique identification code that corresponds to the randomization list, ensuring proper allocation without revealing the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm LT4 (Experimental): The intervention will consist of standard treatment with levothyroxine tablets (50ug/day). The treatment will start from the next day after randomization and end at the day of delivery.
  Interventions: Drug: Levothyroxin
- Arm Placebo (Placebo Comparator): The intervention will consist of standard treatment with levothyroxine placebo daily. The treatment will start from the next day after randomization and end at the day of delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxin — Levothyroxin 50ug/d from randomization until delivery
  Arms: Arm LT4
Drug: Placebo — Placebo to levothyroxin
  Arms: Arm Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to evaluate whether levothyroxine supplement improves pregnancy outcomes in women with recurrent pregnancy loss (RPL) and isolated maternal hypothyroidism (IMH).

The main questions it aims to answer are:

Does levothyroxine increase the live birth rate after 24 weeks of gestation? Does levothyroxine improve secondary outcomes such as ongoing pregnancy rates, reduce the incidence of pregnancy loss, or influence maternal and neonatal complications?

Researchers will:

Compare the levothyroxine treatment group (50 µg/day) to the placebo group to assess the impact of the intervention on live birth rates and other pregnancy outcomes.

Participants will:

Be randomly assigned to receive either levothyroxine or a placebo. Take the assigned treatment daily starting from enrollment until the end of pregnancy.

Undergo routine follow-up visits to monitor pregnancy progress and outcomes. This trial seeks to determine whether routine levothyroxine supplementation can improve pregnancy outcomes for women with RPL and IMH.

DETAILED DESCRIPTION:
Investigators will perform a multi-center, randomized, placebo, double-blind clinical trial of levothyroxine (LT4) in patients aged between 18 years and 40 yearls who are diagnosed with isolated hypothyroxemia (defined as lower FT4 level with normal TSH) and have a previous history of recurrent miscarriages (defined as two or more pregnancy loss). Investigators will assess the effects of standard dose of 50ug/d levothyroxine therapy from the day after randomization to the day of delivery on the pregnancy outcomes, including live birth, neonatal complications, and adverse pregnancy outcomes, etc.

ELIGIBILITY:
Inclusion Criteria:

* women with singleton pregnancy
* women with a history of recurrent pregnancy loss (defined as two or more pregnancy loss before 20wks)
* women diagnosed with isolated maternal hypothyroidism (defined as isolated lower level of FT4 with normal TSH levels) in the current pregnancy before 20wks

Exclusion Criteria:

* patients with known thyroid disorders
* patients with antiphospholipid syndrome or other autoimmune conditions
* patients with contraindications to levothyroxine (e.g., acute cardiac arrest, acute pancreatitis, acute myocarditis)
* patients attending other ongoing clinical trials or unwilling to participate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with confirmed pregnancy
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Live birth after 28 weeks of gestation | From the enrollment to the day of delivery after 28+0 weeks of gestation
  Live birth following spontaneous labor or iatrogenic delivery after 28+0 weeks of gestation (196 days from the participant's last menstrual period)

SECONDARY OUTCOMES:
Ongoing pregnancy at 7 weeks of gestation | From the day of randomization to the 7 weeks of gestation
  ultrasound diagnosis of ongoing pregnancy at 7 weeks of gestation
Ongoing pregnancy at 12 weeks of gestation | From the day of randomization to the 12 weeks of gestation
  ultrasound diagnosis of ongoing pregnancy at 12 weeks of gestation
Ongoing pregnancy at 24 weeks of gestation | From the day of randomization to the 24 weeks of gestation
  ultrasound diagnosis of ongoing pregnancy at 24 weeks of gestation
Miscarriage | From enrollment to 19+6 weeks of gestation
  pregnancy loss before 20 weeks of gestation
Stillbirth | From enrollment to the day of delivery of the dead fetus from 20+0 weeks onward
  fetal death delivered beyond 20 weeks of gestation
Ectopic pregnancy | From enrollment to the end of treatment up to 20 weeks
  ultrasound diagnosis of ectopic pregnancy
Abortion | From enrollment to the day of termination of pregnancy up to 27+6 weeks
  personal request the termination of pregnancy without medical conditions
Need for cervical cerclage | From enrollment to the day of cervical cerlage performed up to 27+6 weeks
  medically indicated cervical cerclage up to 27+6 weeks of gestation
Preterm birth | From enrollment to the day of preterm birth between 28+0 and 36+6 weeks
  live birth between 28+0 and 36+6 weeks of gestation
Gestational age at delivery | up to delivery
  Gestational age at delivery
Antepartum complications | From enrollment to the day of delivery, up to 42+0 weeks
  including: preeclampsia, gestational diabetes, fetal growth restriction
Intrapartum complications | up to delivery
  including: fetal distress, dystocia, fever
Postpartum complications | up to 42 days after childbirth
  including: postpartum hemorrhage, infection, fever
Neonatal birthweight | up to delivery
  the birthweight of the neonate: unit (kg)
Neonatal APGAR score | up to 5 minutes after delivery
  Neonatal APGAR score at 1 and 5 minutes
Neonatal complications | up to 7 days after delivery
  include neonatal breathing disorders, neonatal infections, neonatal asphyxia, neonatal jaundice, NICU admission for any other causes

OTHER OUTCOMES:
Adverse outcomes related to levothyroxine treatment | From enrollment to the end of treatment, up to 40 weeks
  unexpected medical event in a patient or clinical trial participant receiving a pharmaceutical product, which may not necessarily be causally related to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Luo, Ph.D., Principal Investigator — luoq@zju.edu.cn
Locations (2):
- China (2):
  - Zhejiang Women's Hospital, Hangzhou, Zhejiang
  - Zhejiang People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data may be made available at reasonable request on the principal investigator.

REFERENCES:
- [Background] Dhillon-Smith RK, Middleton LJ, Sunner KK, Cheed V, Baker K, Farrell-Carver S, Bender-Atik R, Agrawal R, Bhatia K, Edi-Osagie E, Ghobara T, Gupta P, Jurkovic D, Khalaf Y, MacLean M, McCabe C, Mulbagal K, Nunes N, Overton C, Quenby S, Rai R, Raine-Fenning N, Robinson L, Ross J, Sizer A, Small R, Tan A, Underwood M, Kilby MD, Boelaert K, Daniels J, Thangaratinam S, Chan SY, Coomarasamy A. Levothyroxine in Women with Thyroid Peroxidase Antibodies before Conception. N Engl J Med. 2019 Apr 4;380(14):1316-1325. doi: 10.1056/NEJMoa1812537. Epub 2019 Mar 23. PMID 30907987
- [Background] van Dijk MM, Vissenberg R, Fliers E, van der Post JAM, van der Hoorn MP, de Weerd S, Kuchenbecker WK, Hoek A, Sikkema JM, Verhoeve HR, Broeze KA, de Koning CH, Verpoest W, Christiansen OB, Koks C, de Bruin JP, Papatsonis DNM, Torrance H, van Wely M, Bisschop PH, Goddijn M. Levothyroxine in euthyroid thyroid peroxidase antibody positive women with recurrent pregnancy loss (T4LIFE trial): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2022 May;10(5):322-329. doi: 10.1016/S2213-8587(22)00045-6. Epub 2022 Mar 14. PMID 35298917